CLINICAL TRIAL: NCT02395718
Title: Acute Medical Admission of ELDERly Patients (≥75yrs) to Either Fast Track or Traditional Inward Hospitalisation. A Randomised Controlled Trial
Brief Title: Acute Medical Admissions of ELDERly Patients (ELDER)
Acronym: ELDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: Region Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ELDER
Record Dates: First submitted 2015-01-07; First posted 2015-03-24 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Geriatric Disorder
Keywords: elderly; quick diagnostic unit; short stay unit; randomised controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QDU (Experimental): Patients will undergo a fast track model for diagnostics and treatment with a goal of accomplishing a short-term hospitalisation. Patients will have immediate access to all diagnostic tests and treatments that will be carried out all day (24 hours) on demand from the responsible physician. The QDU is both organisationally and physically integrated in the ED. Point of care ultrasonography can be performed round the clock. Additionally the Department of Radiology provides the QDU with more advanced diagnostic procedures such as e.g. CT scans or MRI scans on a fast track basis. There is access to additional specialist evaluations from the ED staff or from various in house specialists, when needed. Simultaneously to the medical treatment, physical therapists and occupational therapists train and optimise patients' level of functioning, including prevention of loss of function.
  Interventions: Other: QDU
- DIM (Active Comparator): Patients in the control group are treated as conventionally at one of seven wards at the DIM. After initial admission including initial diagnostics and treatment have been carried out in the ED, patients are transferred to the DIM. Usually patients are seen primarily by the on-call physician for evaluation of acute symptoms. The following day, a Chief physician will work out a plan for further diagnostics and treatment. Treatment by physiotherapists and occupational therapists is available on request from a physician. Analyses of blood samples are performed at the central laboratory and radiological procedures at the Department of Radiology.
  Interventions: Other: DIM

INTERVENTIONS:
Other: QDU — Treatment in a QDU. Intervention being fast track model for diagnostics and treatment with a goal of accomplishing a short-term hospitalisation (see description QDU arm)
  Arms: QDU
Other: DIM — Treatment at a ward at the DIM. Traditional inward hospitalisation
  Arms: DIM

SUMMARY:
To evaluate differences in health outcomes among elderly patients (age ≥ 75 years) treated in a Quick Diagnostic Unit (QDU) compared to the Department of Internal Medicine (DIM). A QDU is a medical Short Stay Unit (SSU).

DETAILED DESCRIPTION:
The Danish emergency care system is undergoing major changes; Emergency Departments (ED) are now centralised at fewer hospitals, thus the ED now serve as the single point of entry for all acute patients. Another initiative, has been the establishment of a Quick Diagnostic Unit (QDU) as a subunit in the ED. The QDU is a ward for fast track diagnostics and treatment of stable medical patients that is believed to optimise in-hospital care by quicker diagnosis and shorter hospitalisations, and minimise time for patients to return to their habitual health status. However, little evidence exists on the putative benefits for elderly patients treated in a QDU setting.

In this study, we will examine the benefits and drawbacks of treatment of elderly medical patients (≥75 years) in an acute treatment system with the possibility of fast-track admission and treatment, rather than treatment in the traditional medical system. We will randomise patients to treatment in either a fast track ward/short stay unit, the QDU, or to standard treatment at the Dept. of Internal Medicine (DIM).

We hypothesise that treatment in a QDU compared to DIM offers optimised care through immediate access to clinical staff and rapid diagnostic facilities, treatment and quicker rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 75 years
2. Admitted for in-hospital treatment for an internal medicine disease
3. Green tag triaged upon arrival in the ED

Exclusion Criteria:

1. Previous participation in this trial
2. Participation in other clinical trials
3. No QDU beds available
4. Subject does not have a Danish Civil Registration Number (CPR).
5. Subject resides abroad
6. Requires help using the toilet in daily life
7. Patients not aware of date, time and location, or their own data (name, birth date)
8. Informed consent cannot be obtained

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 430 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 90 days
  Number of participants that die by any cause within 90 days after the day of admission, data will be retrieved from The Danish Civil Registration system 90 days after admission. Accounted as dead or alive.

SECONDARY OUTCOMES:
Length of stay in-hospital | Lenght of stay is assessed from date of randomization untill the date of discharge, date of death from any cause or whichever came first, assessed up to 100 weeks.
  Length of stay in-hospital per participant, defined as the duration of a single episode of hospitalisation including day of admission, and day of discharge. Length of stay will be calculated by subtracting the day of admission from day of discharge as registered in the patient's hospital chart. Accounted in days
Readmissions | 30 days
  Number of participants that are readmitted within 30 days from date of discharge (defined as the proportion of patients readmitted no more than 30 days post initial discharge as registered in the patient's hospital chart. Accounted as yes or no).
In hospital Mortality | In hospital mortality is assessed from date of randomization untill the date of discharge, date of death from any cause or whichever came first, assessed up to 100 weeks.
  Number of participants that die In-hospital (defined as patients that have died at any time during hospitalisation as registered in the patient's hospital chart. Accounted as dead or alive).
In-hospital Transfer | is assessed from date of randomization untill the date of discharge, date of death from any cause or whichever came first, assessed up to 100 weeks.
  Number of participants that are transferred to other wards while in hospital (defined as patients that have been transferred to any other ward in the hospital apart from the Department of Radiology at any time during hospitalisation as registered in the patient's hospital chart. Accounted as yes or no).
Instrumental Activities of Daily Living | 90 days (± 2 days) from date of randomization
  Number of participants with change in Instrumental activities of daily living-score (iADL- score) within 90 days from admission (defined as any decrease or increase in iADL score within 90 days from admission. Accounted in score increase, score decrease or no-change).
Placement in a long-term-care home after hospitalisation. | 3 months (± 2 days)
  Number of participants that are placed in a long-term-care home after hospitalisation within 90 days from admission (defined by placement in any kind of long-term-care home after hospitalisation from the first day of admission to day 90 after admission. Accounted as yes or no).
Complications of hospitalisation | is assessed from date of randomization untill the date of discharge, date of death from any cause or whichever came first, assessed up to 100 weeks.
  Number of participants with complications of hospitalisation (defined as an injury caused by medical management (rather than the disease process).
  Complications of hospitalisation are one or more of the following:
  1. Nosocomial infection
  2. Medication error
  3. Deep venous thrombosis
  4. Pulmonary Embolism
  5. Delirium
  6. Decubitus ulcers
  7. Post-procedural haemorrhage
  8. In-hospital fractures or falls
  9. Gastrointestinal haemorrhage
  10. Cerebral infarction

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Stroem, MD, Principal Investigator — Dept. of Emergency Medicine, Holbaek Sygehus, Copenhagen University Hospital
Locations (1):
- Dept. of Emergency Medicine, Holbaek Sygehus, Copenhagen University Hospital, Holbæk, Denmark

REFERENCES:
- [Derived] Strom C, Rasmussen LS, Lowe AS, Lorentzen AK, Lohse N, Madsen KHB, Rasmussen SW, Schmidt TA. Short-stay unit hospitalisation vs. standard care outcomes in older internal medicine patients-a randomised clinical trial. Age Ageing. 2018 Nov 1;47(6):810-817. doi: 10.1093/ageing/afy090. PMID 29905758
- [Derived] Strom C, Rasmussen LS, Wistisen Rasmussen S, Benn Madsen KH, Ancher Sorensen HA, Andersen Schmidt T. Admission of elderly medical patients to fast track or standard hospitalisation: protocol for a randomised trial. Dan Med J. 2016 Mar;63(3):A5189. PMID 26931195